CLINICAL TRIAL: NCT03175900
Title: Effectiveness and Neural Mechanism of Naoan Dripping Pills for Migraine: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effectiveness and Neural Mechanism of Naoan Dripping Pills for Migraine
Acronym: ENMNM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Zhejiang Liaoyuan Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Ying Gao, Vice president of Dongzhimen Hospital, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-2016-84-01
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Migraine
Keywords: Migraine; Naoan dripping pills; Traditional Chinese Medicine; fMRI; Randomized Controlled trial
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naoan dripping pills for migraine (Experimental): Drug: Naoan dripping pills, Chinese patent medicine，pill. Patients will receive treatment with Naoan dripping pills for 12 weeks, Fenbid can be taken if headache is unbearable Procedure: MRI scanning（fMRI and DTI）
  Interventions: Drug: Naoan dripping pills
- Placebo (Placebo Comparator): Drug: Placebo, pill. Patients will receive treatment with placebo for 12 weeks, Fenbid can be taken if headache is unbearable Procedure: MRI scanning （fMRI and DTI）
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naoan dripping pills — Patients will take 20 pills(1000mg) after meal twice a day for 12 weeks, Fenbid can be taken if headache is unbearable, but make sure the records(including attack time, drug dosage, pain intensity and duration) are written down as detailed as possible.
  Procedure: MRI scanning (fMRI and DTI）
  Arms: Naoan dripping pills for migraine
Drug: Placebo — Patients will take 20 pills(1000mg) after meal twice a day for 12 weeks, Fenbid can be taken if headache is unbearable, but make sure the records(including attack time, drug dosage, pain intensity and duration) are written down as detailed as possible.
  Procedure: MRI scanning (fMRI and DTI)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial. Its main purpose is to investigate the effects and neural mechanism of Naoan dripping pills on migraine patients by utilizing fMRI and DTI method, as well as headache evaluation measures such as responder rate, headache duration, PRO scale, etc.

DETAILED DESCRIPTION:
Naoan dripping pills, which is a Chinese patent medicine proved effectively in treating migraine on clinic, but its neural mechanism remains unknown. This study is expected to validate the effectiveness and explore its neural mechanism by fMRI and DTI so as to provide evidence for physicians to promote the appropriate use of Naoan dripping pills treatment for migraine patients. Patients will be randomly assigned to either Naoan dripping pills group or placebo group, they will receive Naoan dripping pills/Placebo treatment for 12 weeks. Clinical evaluation will be performed at baseline, every 4 weeks during treatment and the follow-up week(16 weeks) . MRI scans are performed at baseline, and 12 weeks later. Responder rate (defined as the percentage of subjects in a treatment group with 50 % or greater reduction in attack frequency during treatment compared with the baseline period) and fMRI and DTI imaging changes after treatment are defined as primary outcome. In addition, 10 healthy controls will also undergo MRI scanning at baseline to determine abnormal brain activity and structure in migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has migraine without aura or with typical aura according to criteria of the International Headache Society (IHS)
* Subject has been diagnosed with qi deficiency syndrome and/or blood stasis syndrome in TCM
* Subject has onset of migraine occurring before age 50
* Subject has a history of migraine headaches for at least 1 year
* In recent 3 months, subject has 2 to 8 headache attacks every 4 weeks
* Age ≥ 18 years and ≤ 65 years
* Right-handers
* Subject has signed informed consent

Exclusion Criteria:

* Subject takes painkillers more than 10 days a month for headache attacks
* Subject who was／is in possess of Naoan dripping pills therapy but the treatment is ineffective
* Allergic to Naoan dripping pills
* subject's taken, within 12 weeks before enrollment, migraine prevention drugs drugs such as β-blocker, calcium channel inhibitor，Anti-epileptic drugs，antidepressants or 5-HT receptor blocker
* Alcohol or drug abusers
* Subject suffers from other primary headaches as specified by IHS criteria
* Subject has medical condition such as severe heart disease, stroke, kidney disease, liver disease, hepatic or renal impairment, hematologic disease
* Subject has psychological or mental disorder, Hamilton Anxiety Scale（HAMA）≥7，Hamilton Depression Scale（HAMD）≥7
* Subject has language impairment or cognitive impairment, unable to read, understand or record information in study diaries and questionnaires
* Pregnant or breast feeding subjects
* Subjects with contraindications for undergoing MRI scans (e.g. Claustrophobic, patients with heart pacemaker )

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-08-04 (Actual)

PRIMARY OUTCOMES:
Responder rate | 12 weeks
  Defined as the percentage of subjects in a treatment group with 50 % or greater reduction in attack frequency during treatment compared with the baseline period

SECONDARY OUTCOMES:
Change in functional connectivity assessed by Resting-state fMRI | Baseline and 12 weeks
  Investigate the differences in fractional anisotropy of migraine patients compared to healthy volunteers at baseline, and compare the changes of fractional anisotropy after 12 weeks' treatment in two groups
Change in fractional anisotropy (FA) assessed by DTI | Baseline and 12 weeks
  Investigate the differences in fractional anisotropy of migraine patients compared to healthy volunteers at baseline, and compare the changes of fractional anisotropy after 12 weeks' treatment in two groups
Duration of migraine attacks | 12 weeks and 16 weeks
  To compare the reduction of duration of migraine attacks after 12 weeks' treatment in two groups
Intensity of headache | 12 weeks and 16 weeks
  To compare the change of the duration of migraine attacks (mild, moderate, severe) after 12 weeks' treatment in two groups
Patient reported outcome (PRO) scale of migraine | 12 weeks and 16 weeks
  To compare the change of Patient reported scores after 12 weeks' treatment in two groups
Number of migraine days per evaluation interval | 12 weeks and 16 weeks
  To compare the reduction of the number of migraine days per evaluation interval after 12 weeks' treatment in two groups
Drug consumption for symptomatic or acute treatment | 12 weeks and 16 weeks
  To compare the change of drug consumption for symptomatic or acute treatment after 12 weeks' treatment in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No